CLINICAL TRIAL: NCT07014189
Title: Open-label Multicenter Non-inferiority Trial of Nevirapine Plus Lamivudine Versus Optimal Standard in HIV Maintenance Therapy
Brief Title: Nevirapine / Lamivudine for HIV Maintenance Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Christian R Kahlert, MD, principal investigator, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU 17/027
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection; Antiretroviral Treatment; Maintenance Therapy
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Active Comparator): Lamivudin / Nevirapine
  Interventions: Drug: Neviparine (NVP)/ Lamivudine (3TC)

INTERVENTIONS:
Drug: Neviparine (NVP)/ Lamivudine (3TC) — Treatment with nevirapine (400mg retard) and lamivudine (300mg) once daily

SUMMARY:
The standard treatment for HIV infection involves taking a combination of three HIV drugs. The main reason for using multiple substances is to prevent resistance from developing rapidly when only one or two drugs are used.

However, in recent years, studies have shown that the risk of resistance developing is significantly lower once viral replication in the body has been completely suppressed. Studies have now been conducted on this maintenance therapy phase, which aims to reduce the number of drugs used.

Some positive results have been reported with monotherapy. There have been positive results with both protease and integrase inhibitors. However, both groups of drugs demonstrate monotherapy failure in 10-20% of patients. We suspect that poor penetration into the genital tract and brain is partly responsible for this.

In contrast, recent studies on the dual combination of protease or integrase inhibitors with lamivudine have demonstrated excellent efficacy. Lamivudine is known to work very well in the brain and genital tract. Since HIV medication must be taken for life, simplifying therapy is very important. This reduces the potential for long-term side effects and costs.

The Clinic for Infectious Diseases and Hospital Hygiene at the Cantonal Hospital of St. Gallen in Switzerland has many years of experience with nevirapine, an HIV medication introduced over 20 years ago. One third of patients are treated with this substance. Of the additional preparations used in combination with nevirapine, one contains lamivudine (or its analogue, emtricitabine), plus either abacavir or tenofovir. The latter two have potentially significant long-term side effects, including an increased risk of cardiovascular disease and kidney/bone toxicity.

A dual combination of nevirapine and lamivudine is highly likely to be effective. Furthermore, it is the most favourable of all the alternative combinations. Based on current knowledge, this combination appears to have no long-term side effects.

After conducting a controlled pilot study with 20 patients at the KSSG (Kahlert, 2020, https://doi.org/10.1371/journal.pone.0237770), data was obtained showing that the combination of nevirapine and lamivudine is effective in maintaining viral suppression. None of the patients experienced 'viral blips' (temporarily detectable virus concentrations of 50-200 HIV RNA copies/ml of blood), which are known to occur in monotherapy studies. After an observation period of 72-96 weeks, all patients showed sustained stable viral suppression (<50 HIV RNA copies/ml of blood).

The aim of this study is to evaluate the dual combination of nevirapine and lamivudine in a multicentre setting. The intervention involves switching well-selected patients with no history of treatment failure who have been on long-term, stable, well-suppressed HIV therapy with nevirapine from triple combination therapy to nevirapine plus lamivudine. The study is a non-inferiority trial compared to a virtual control group receiving stable standard combination therapy with 0% treatment failure.

The primary outcome parameter used to assess the non-inferiority of the dual combination is the proportion of patients experiencing treatment failure, as determined by a viral load of ≥200 HIV RNA copies/ml at weeks 6, 12, 24, 36 and 48 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients on a stable HIV-therapy containing NVP for at least six months
* Duration of viral load suppression (HIV-RNA < 50 cp/ml) of more than 2 years (allowing occasional blips, i.e. viral load measurements of 50-200 HIV-RNA cp/ml followed by an additional measurement of <50 cp/ml within 4 weeks)
* No previous failure of any NNRTI based therapy
* No known resistance to NVP or 3TC
* Able to fully understand the informed consent and the experimental nature of the study
* Absence of any health believe systems that might interfere with drug intake

Exclusion Criteria:

* Chronic hepatitis B infection (HBs-AG positive)
* Any condition, that might, at the discretion of the principle investigator, interfere with treatment adherence or regular HIV-RNA testing appointments, such as i) psychiatric disorders, ii) known adherence problems in the past 2 years or iii) health believe issues known to cause patients to stop treatment (e.g. expecting God to cure HIV or not believing the existence of HIV, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV-RNA ≥ 200 cp/ml | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Vernazza, Professor, Study Director — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
decision will be taken, when there is a reasonable request for the data